CLINICAL TRIAL: NCT06745323
Title: A Phase 2, Open-label, Randomized, Multicenter Study of Tarlatamab Dosing Regimens in Subjects With Small Cell Lung Cancer (SCLC) (DeLLphi-309)
Brief Title: A Phase 2, Open-label, Randomized, Multicenter Study of Tarlatamab Dosing Regimens in Subjects With SCLC
Acronym: DeLLphi-309
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240092
Expanded Access: Available
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Small Cell Lung Cancer (SCLC)
Keywords: Tarlatamab; AMG 757
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — AMG 757

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Arm A: Dose 1 Tarlatamab (Experimental): Participants will receive dose 1 of Tarlatamab by intravenous (IV) infusion during the treatment period.
  Interventions: Drug: Tarlatamab
- Treatment Arm B: Dose 2 Tarlatamab (Experimental): Participants will receive dose 2 of Tarlatamab by IV infusion during the treatment period.
  Interventions: Drug: Tarlatamab
- Treatment Arm C: Dose 3 Tarlatamab (Experimental): Participants will receive dose 3 of Tarlatamab by IV infusion during the treatment period.
  Interventions: Drug: Tarlatamab

INTERVENTIONS:
Drug: Tarlatamab — Tarlatamab will be administered by IV infusion.
  Other Names: AMG 757

SUMMARY:
The primary objective of this study is to describe the antitumor activity of tarlatamab in participants with small cell lung cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent prior to initiation of any study specific activities/procedures.
* Age ≥ 18 years (or legal adult age within country, whichever is older) at the time of signing the informed consent.
* Histologically or cytologically confirmed SCLC with demonstrated progression or relapse.
* Participants who progressed or recurred following 1 platinum-based regimen.
* Measurable disease as defined per RECIST 1.1 within the 21-day screening period.
* Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1.
* Minimum life expectancy of 12 weeks.
* Adequate organ function as described per protocol.

Exclusion Criteria:

* Disease Related

  * Previous diagnosis of transformed non-small cell lung cancer (NSCLC) including epidermal growth factor receptor activating mutation positive NSCLC that has transformed to SCLC.
  * Symptomatic central nervous system (CNS) metastases with exceptions defined in the protocol.
* Other Medical Conditions

  * History of other malignancy within the past 2 years, with exceptions defined in the protocol.
  * Evidence of interstitial lung disease or active, non-infectious pneumonitis
  * Diagnosis or evidence of leptomeningeal disease.
  * Active autoimmune disease that has required systemic treatment (except replacement therapy) within the past 2 years or any other diseases requiring immunosuppressive therapy while on study.
  * History of solid organ transplantation.
  * Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association > class II) within 6 months prior to first dose of study treatment.
  * History of arterial thrombosis (eg, stroke or transient ischemic attack) within 6 months prior to first dose of study treatment
  * Presence or history of viral infection based on criteria per protocol.
  * Symptoms and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection requiring antibiotics within 7 days prior to the first dose study treatment.
  * Known or active infection requiring parenteral antibiotic treatment.
  * History of severe or life-threatening events from any immune-mediated therapy.
  * Major surgical procedures within 21 days of prior to first dose of study treatment.
* Prior/Concomitant Therapy

  * Prior anticancer therapy within 30 days of enrollment (14 days for conventional chemotherapy).
  * Prior enrollment on a tarlatamab clinical trial OR prior therapy with any selective inhibitor of the DLL3 pathway.
  * Current anti-cancer therapy such as chemotherapy, immunotherapy, or targeted therapy with exceptions.
  * Receiving systemic corticosteroid therapy or any other immunosuppressive therapy within 7 days prior to first dose as described per protocol.
  * Live and live-attenuated vaccines within 14 days prior to the start of study treatment. Inactive vaccines and live viral non-replicating vaccines within 3 days prior to the first dose of study treatment.
* Prior/Concurrent Clinical Study Experience

  * Currently receiving treatment in another investigational device or drug study, or less than 30 days or 5 half-lives since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Other Exclusions

  * Female participants of childbearing potential unwilling to use protocol specified method of contraception during treatment and for an additional 60 days after the last dose of tarlatamab.
  * Female participants who are breastfeeding or who plan to breastfeed while on study through 60 days after the last dose of tarlatamab.
  * Female participants planning to become pregnant or donate eggs while on study through 60 days after the last dose of tarlatamab.
  * Female participants of childbearing potential with a positive pregnancy test assessed at screening and/or day 1 by a highly sensitive urine or serum pregnancy test.
  * Male participants with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 60 days after the last dose of tarlatamab.
  * Male participants with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for an additional 60 days after the last dose of tarlatamab.
  * Male participants unwilling to abstain from donating sperm during treatment and for an additional 60 days after the last dose of tarlatamab.
  * Participant has known sensitivity or is contraindicated to any of the products or components to be administered during dosing.
  * Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures.
  * History or evidence of any other clinically significant disorder, condition or disease determined by the investigator or Amgen physician, if consulted, would pose a risk to the subject safety or interfere with the study evaluation procedure or completion.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2029-02-13 (Estimated); Study Completion 2029-02-13 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with confirmed objective response to Tarlatamab | Approximately 52 Months
Proportion of participants with complete response to Tarlatamab | Approximately 52 Months
Proportion of participants with partial response to Tarlatamab | Approximately 52 Months

SECONDARY OUTCOMES:
Average serum concentrations of Tarlatamab | Approximately 52 Weeks
Duration of confirmed response, defined as the time from the first documentation of OR until the first documentation of disease progression or death | Approximately 52 Months
Disease control, defined as objective response or stable disease | Approximately 52 Months
Duration of disease control | Approximately 52 Months
Progression-free survival, defined as the time from randomization to the first documentation of disease progression or death due to any cause | Approximately 52 Months
Objective response, defined as best overall response of CR or PR | Approximately 52 Months
Overall survival, defined as the time from randomization to death due to any cause | Approximately 52 Months
Overall Survival rate at 6 months and 1 year from randomization | Approximately 52 Months
Number of participants with treatment-emergent adverse events | Approximately 52 Months
Number of participants with anti-tarlatamab antibody formation | Approximately 52 Months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (78):
- United States (12):
  - University of California Los Angeles, Los Angeles, California
  - Hartford HealthCare Cancer Institute at The Hospital of Central Connecticut, Plainville, Connecticut
  - AdventHealth Hematology and Oncology, Orlando, Florida
  - City of Hope Chicago, Rockford, Illinois
  - Health Partners Cancer Center at Regions Hospital, Saint Paul, Minnesota
  - New York Oncology Hematology PC, Albany, New York
  - Duke University, Durham, North Carolina
  - FirstHealth Cancer Center, Pinehurst, North Carolina
  - Guthrie Medical Group, Sayre, Pennsylvania
  - Tennessee Oncology PLLC - Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Virginia Cancer Specialists PC, Fairfax, Virginia
- Argentina (2):
  - Fundacion Respirar, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones clinicas de Mar del Plata, Mar del Plata, Buenos Aires
- Australia (2):
  - Monash Medical Centre, Clayton, Victoria
  - Austin Health, Austin Hospital, Heidelberg, Victoria
- Belgium (3):
  - Grand Hopital de Charleroi - Site des Viviers, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
- Brazil (6):
  - Liga Norte-Riograndense Contra O Cancer, Natal, Rio Grande do Norte
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Cipo - Centro Integrado de Pesquisa em Oncologia, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor, Barretos, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
- China (12):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
- France (3):
  - Hopital Lyon sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Hopital Foch, Suresnes
- Germany (4):
  - Helios Kliniken Emil-von-Behring, Berlin
  - Universitaetsklinikum des Saarlandes, Homburg
  - Universitaetsklinikum Schleswig-Holstein - Kiel, Kiel
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (6):
  - Henry Dunant Hospital Center, Athens
  - Alexandra Hospital, Athens
  - Metropolitan Hospital, Athens
  - University Hospital of Heraklion, Heraklion - Crete
  - University Hospital of Patras, Pátrai
  - European Interbalkan Medical Center, Thessaloniki
- Azienda Ospedaliera San Giovanni Addolorata, Roma, Italy
- Japan (8):
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kanagawa Prefectural Hospital Organization Kanagawa Cancer Center, Yokohama, Kanagawa
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju Chungbuk
  - Kyungpook National University Chilgok Hospital, Daegu
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Severance Hospital Yonsei University Health System, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (5):
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Complexo Hospitalario Universitario A Coruna Hospital Teresa Herrera, A Coruña, Galicia
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (2):
  - Kantonsspital Baden, Baden
  - Universitaetsspital Zuerich, Zurich
- Turkey (Türkiye) (5):
  - Baskent Universitesi Adana Doktor Turgut Noyan Uygulama ve Arastirma Merkezi, Adana
  - Memorial Ankara Hastanesi, Ankara
  - Gazi Universitesi Saglik Arastirma ve Uygulama Merkezi Gazi Hastanesi, Ankara
  - Goztepe Prof Dr Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
- Christie Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com